CLINICAL TRIAL: NCT07221695
Title: Foam Plus Glue Versus Foam Plus Coils for Ovarian Vein Embolization in the Treatment of Pelvic Venous Disorders:
Brief Title: Embolization Strategies for Pelvic Venous Disorders: Foam + Glue vs Foam + Coils
Acronym: foam and coil
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Moustafa Hassan Mabrouk Abdelhameed, principal investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: glue vs coil for ovarian ttt
Record Dates: First submitted 2025-10-12; First posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Pelvic Congestive Syndrome
MeSH Terms: interventions — Enbucrilate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Embolization using polidocanol foam followed by N-butyl cyanoacrylate (Active Comparator): . After selective catheterization of the ovarian vein and reflux confirmation, Sclerosant foam will be prepared using 3% polidocanol (Aethoxysklerol®, Kreussler Pharma), mixed with room air in a 1:4 ratio (1 mL polidocanol to 4 mL air) using the Tessari double-syringe technique, creating a dense and stable foam. The foam will be injected slowly into the reservoir of the refluxing segment of the ovarian vein under fluoroscopic guidance to induce endothelial irritation and reduce venous flow. A total of 5-10 mL of 3% polidocanol foam will be injected per vein, adjusted based on vein diameter and reflux length.
  Next, N-butyl cyanoacrylate (Gluebran®️ 2) will be mixed with Lipiodol in a 1:2 to 1:3 ratio, depending on vein size and flow rate. Approximately 1-2 mL of the glue mixture will be injected per vein using a coaxial microcatheter system from distal to proximal segments. Occlusion will be confirmed by post-embolization venography."
  Interventions: Other: Foam + N-butyl Cyanoacrylate
- Combined Foam Sclerotherapy and Detachable Coil Embolization (Active Comparator): Patients in this group will undergo embolization using sclerosant foam followed by detachable platinum coils. Vascular access and catheterization technique will mirror Group A.
  After injecting polidocanol foam (as above), subsequently, detachable platinum fibered coils - specifically Interlock™ (Boston Scientific) or Concerto™ (Medtronic) - will be deployed to achieve permanent mechanical occlusion. Coil selection (diameter and length) will be based on intra-procedural vein sizing. Final occlusion will be confirmed via completion venography.
  Interventions: Other: Combined Foam Sclerotherapy and Detachable Coil Embolization

INTERVENTIONS:
Other: Foam + N-butyl Cyanoacrylate — 3% polidocanol (Aethoxysklerol®, Kreussler Pharma), mixed with room air in a 1:4 ratio (1 mL polidocanol to 4 mL air) using the Tessari double-syringe technique, creating a dense and stable foam.
  Arms: Embolization using polidocanol foam followed by N-butyl cyanoacrylate
Other: Combined Foam Sclerotherapy and Detachable Coil Embolization — polidocanol foam (as above), subsequently, detachable platinum fibered coils - specifically Interlock™ (Boston Scientific) or Concerto™ (Medtronic)
  Arms: Combined Foam Sclerotherapy and Detachable Coil Embolization

SUMMARY:
Foam Plus Glue Versus Foam Plus Coils for Ovarian Vein Embolization in the Treatment of Pelvic Venous Disorders: A Randomized Controlled Trial

ELIGIBILITY:
Inclusion Criteria

* Female patients aged 18 to 50 years
* Clinically suspected pelvic venous disorder (PVD), presenting with chronic pelvic pain ≥ 6 months
* Pelvic pain intensity ≥ 4 on a 10-point Visual Analogue Scale (VAS) at baseline
* No evidence of significant venous obstruction or internal iliac insufficiency
* Willingness to participate, provide written informed consent, and comply with study visits and procedures exclusion criteria
* Pregnancy or planning to conceive within the next 12 months
* Significant Nutcracker syndrome diagnosed by duplex / CTV / MRV
* Significant May-Thurner syndrome diagnosed by duplex / CTV / MRV
* Non-ovarian sources of reflux requiring intervention, including internal iliac vein insufficiency; During venography all patients will undergo selective pelvic venography prior embolization to exclude patients who have combined gonadal and internal iliac vein reflux)
* History of previous pelvic vein embolization or surgical ligation
* Coagulopathy, defined as:

  * INR > 1.5
  * Platelet count < 50 × 10⁹/L
* Severe comorbidities, including:

  * Active pelvic infection (e.g., pelvic inflammatory disease)
  * End-stage renal disease (eGFR < 30 mL/min/1.73 m²)
  * Decompensated heart failure (NYHA class III-IV)
  * Active malignancy requiring treatment

Known allergy or hypersensitivity to:

* Iodinated contrast media
* Polidocanol (Aethoxysklerol®)
* N-butyl cyanoacrylate (e.g., Gluebran® 2)
* Nickel, platinum, or stainless steel (components of embolization coils) . Presence of non-venous pelvic pathology requiring immediate management

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
compare the clinical efficacy of ovarian vein embolization using combined foam plus N-butyl cyanoacrylate (Gluebran®️) versus combined foam plus detachable coils | 18 months
  2. Symptom severity reduction, assessed by the Pelvic Venous Clinical Severity Score (PVCSS) at baseline, 3, 6, 12, and 18 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr El Shaykh University, Kafr ash Shaykh, Kafrelshaykh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes